CLINICAL TRIAL: NCT05518877
Title: Low Dose Ketamine Infusion for Analgesia in the Emergency Department (ED) to Reduce Side Effects: A Double Blind, Double Dummy Randomized Controlled Trial
Brief Title: Low Dose Ketamine Infusion for Analgesia in the Emergency Department to Reduce Side Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22194
Record Dates: First submitted 2022-04-15; First posted 2022-08-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pain, Acute; Dissociation
MeSH Terms: conditions — Acute Pain; Dissociative Disorders | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Double-blind, double-dummy randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine 15 Minutes (Active Comparator): Participants receive 0.25mg/kg Ketamine dose intravenous for pain over 15 minutes.
  Interventions: Drug: Ketamine
- Ketamine 30 Minutes (Experimental): Participants receive 0.25mg/kg Ketamine dose intravenous for pain over 30 minutes.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Administration of Ketamine
  Other Names: Ketalar

SUMMARY:
This will be an intent to treat prospective, double blind, double-dummy, randomized trial. Our primary objective is the reduction of side effects of sub dissociative dose ketamine given by slow intravenous (IV) infusion over 30 minutes vs. 15 minutes in the treatment of acute, severe pain in Emergency Department (ED) patients. The secondary objective will be to maintain adequate pain control (as defined by a Visual Analog Scale (VAS) score of ≤ 5cm) at 30 minutes for both groups.

DETAILED DESCRIPTION:
Previous research has shown that low dose ketamine (LDK) Intravenous push (IVP) (0.3mg/kg) to have equivalent pain reduction in moderate to severe acute pain in the Emergency Department (ED) when compared to standard of care of morphine intravenous push (IVP) (0.1mg/kg). Ketamine has been shown to produce side effects in these studies, including dizziness, feeling of unreality and mood changes, but no unexpected side effects or adverse events. Additional studies have compared IVP with slower infusion of low dose ketamine (LDK) and have shown a decrease in side effects while maintaining similar analgesic efficacy. This previous trial found increased feelings of unreality for the IVP group (difference of 37.5%) as well as increased rates of sedation.

In clinical practice, increasing the time/duration of the infusion has resulted in a decrease of reported side effects from patients while still maintaining analgesia. There have been no studies done to prove that there is a further reduction in side effects with a longer LDK infusion. The investigators believe that increasing the infusion time to greater than 15 minutes will reduce the frequency and intensity of expected side effects of ketamine felt by participants and allow for further use of ketamine as a non-opiate analgesic in the ED.

Overall aims of project:

1. Reduce overall side effects of low dose ketamine when given over 30 minutes versus 15 minutes.
2. Maintain adequate pain control, as defined by a Visual Analogue Scale (VAS) score of ≤5 cm at 30 minutes for both groups.

Hypothesis: Slow infusion of low dose ketamine (LDK) over 30 minutes will provide adequate pain control (as defined by VAS score of ≤5 cm), and reduce incidence and severity (by at least 20% or 1 point on SERSDA scale) of known side effects when compared to LDK given over 15 minutes in moderate to severe acute pain for patients presenting to the ED.

Study Design

The location of this study will be the Akron City Hospital Emergency Department. The trial will enroll approximately 48 participants over a 24-month enrollment period.

This will be an intent to treat prospective, double blind, double-dummy, randomized trial. The primary outcome will be a comparison of side effects of sub dissociative dose ketamine given by slow IV infusion over 15 minutes vs 30 minutes in treatment of moderate to severe acute pain in ED patients. The secondary outcome will be adequate pain control (VAS ≤5 cm), and need for rescue analgesia between the two groups.

The control group will receive slow IV infusion of ketamine over 15 minutes. The experimental group will receive slow IV infusion of ketamine over 30 minutes.

If the potential participant meets all eligibility criteria, they will be consented by study staff members and then randomized to receive Ketamine 0.25mg/kg in 100cc normal saline (NS) as IV infusion over specified time as well as "placebo" 100cc NS over the other time slot.

Pharmacy staff will blind medication as well as provide medication in a blinded fashion to the nurse who will use infusion pumps to deliver both study medication and placebo simultaneously. Nursing staff will receive training on administration of medication prior to starting the study.

The investigators will measure the side effect profile using the Side Effects Rating Scale for Dissociative Anesthetics (SERSDA) along with the VAS (visual analog scale) scores from 0-100mm.

Vital signs (heart rate, blood pressure, respiratory rate and oxygen saturation) will also be obtained at 0, 5, 15, 30, 60, and 90 minutes from the start of the ketamine/NS placebo infusion.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 or older
* Primary complaint of acute moderate to severe pain on VAS/ numeric pain scale (a score of ≥5cm which corresponds to 50mm).
* Pain described as abdominal, flank, back, musculoskeletal, or traumatic chest pain
* Must be alert and oriented times three
* Able to provide consent

Exclusion criteria:

* Pregnant
* Breastfeeding
* Altered mental status
* Known or reported allergy, hypersensitivity or intolerance to ketamine
* Unstable vital signs (systolic blood pressure <80 or >180mmHg, heart rate <50 or >150 beats per minute, and respiratory rate <10 or >30 breaths per minute)
* History of unstable heart disease, such as arrhythmias, congestive heart failure, or coronary heart disease.
* History of untreated or uncontrolled thyroid disease
* Acute head or eye injury
* Active or current use of alcohol or drugs
* Known intracranial hypertension
* Hepatic or renal insufficiency
* Current active manic phase of bipolar disorder
* Active delusions, hallucinations, or schizophrenia
* Patients who have recent fentanyl use within 60 minutes or other analgesic use (opiates) within 4 hours of study enrollment (signing of consent)
* Patients who have enrolled in the study during a previous ED encounter
* Chronic use of opiates (i.e.: fentanyl patch, SR opiates)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) Score | 30 minutes
  Overall side effects as measured by the Side Effect Rating Scale for Dissociative Anesthetics (SERSDA). SERDSA measures severity of nine adverse effects based on a 5-point scale from "0" (no adverse effect) to "4" (very bothersome effect).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Score | 30 minutes
  Severity of Self-Reported Pain on the standard 100mm VAS scale. Visual Analogue Scale scoring is done by asking the subject to mark the spot on the VAS Pain Assessment Tool (0-10cm) to indicate their perception of pain. Following this, the investigator scores the intensity of pain according to the 0-100mm corresponding scale (one instrument i.e., 5cm= 50mm)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pallaci, DO, FACEP, Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884
- [Background] Motov S, Mai M, Pushkar I, Likourezos A, Drapkin J, Yasavolian M, Brady J, Homel P, Fromm C. A prospective randomized, double-dummy trial comparing IV push low dose ketamine to short infusion of low dose ketamine for treatment of pain in the ED. Am J Emerg Med. 2017 Aug;35(8):1095-1100. doi: 10.1016/j.ajem.2017.03.004. Epub 2017 Mar 3. PMID 28283340